CLINICAL TRIAL: NCT02771197
Title: Phase II Trial of Lymphodepletion and Anti-PD-1 Blockade to Reduce Relapse in High Risk AML Patients Who Are Not Eligible for Allogeneic Stem Cell Transplantation
Brief Title: Lymphodepletion and Anti-PD-1 Blockade to Reduce Relapse in AML Patient Not Eligible for Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 1150
Record Dates: First submitted 2016-03-22; First posted 2016-05-13 (Estimated); Results first posted 2023-09-22 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Melphalan; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lymphodepletion plus Pembrolizumab (Experimental): Fludarabine & Melphalan followed by autologous stem cell transplantation. Pembrolizumab will begin on Day +1.
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Fludarabine
Drug: Melphalan
Drug: Pembrolizumab

SUMMARY:
AML is the most common acute leukemia in adults. Most patients can undergo allogeneic stem cell transplantation as a possible cure; however, many patients are not candidates for allogeneic transplant due to age, overall health, psychosocial factors, and/or lack of available donors. Therefore, these patients are unable to receive the therapeutic benefits of the "graft-versus-leukemia" effect of donor immune cells. The aim of this study is to hopefully break immune tolerance to AML cells to provide better outcomes in patients with non-favorable risk AML.

DETAILED DESCRIPTION:
Non-favorable risk AML patients will undergo a preparative regimen of lymphodepletion of Flu/Mel followed by autologous transplantation. Anti-PD-1 therapy of pembrolizumab will begin on Day +1 following stem cell transplantation and will be administered every 3 weeks for a total of 8 doses. According to the literature, the risk of 2-year relapse is estimated to be 60-80% in patients with non-favorable risk AML in CR-1. With this protocol, investigators hypothesize that following lymphodepleting chemotherapy and pembrolizumab, the 2-year relapse risk will decrease to less than or equal to 35%. The one-sided Wald test at 5% significance level will be used to test the hypothesis. The size of 20 patients yields the power of 90.5% assuming that the actual 2-year leukemia-free survival is 60%.

ELIGIBILITY:
Inclusion Criteria:

* Non-favorable risk AML
* In CR-1 or subsequent CR
* Completed at least one cycle of consolidation chemotherapy
* Collection of at least 2x106/kg CD34+ cells
* KPS of 70% or greater

Exclusion Criteria:

* Received investigational agent within 4 weeks of first dose
* Prior chemotherapy, radiation therapy within 2 weeks of first dose
* Hypersensitivity to pembrolizumab or any of its excipients
* Received prior therapy with anti-PD-1, anti-PD-L1, or anti-PD-L2 agent

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Solomon, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (2):
- United States (2):
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cornelissen JJ, van Putten WL, Verdonck LF, Theobald M, Jacky E, Daenen SM, van Marwijk Kooy M, Wijermans P, Schouten H, Huijgens PC, van der Lelie H, Fey M, Ferrant A, Maertens J, Gratwohl A, Lowenberg B. Results of a HOVON/SAKK donor versus no-donor analysis of myeloablative HLA-identical sibling stem cell transplantation in first remission acute myeloid leukemia in young and middle-aged adults: benefits for whom? Blood. 2007 May 1;109(9):3658-66. doi: 10.1182/blood-2006-06-025627. Epub 2007 Jan 9. PMID 17213292
- [Result] Koreth J, Schlenk R, Kopecky KJ, Honda S, Sierra J, Djulbegovic BJ, Wadleigh M, DeAngelo DJ, Stone RM, Sakamaki H, Appelbaum FR, Dohner H, Antin JH, Soiffer RJ, Cutler C. Allogeneic stem cell transplantation for acute myeloid leukemia in first complete remission: systematic review and meta-analysis of prospective clinical trials. JAMA. 2009 Jun 10;301(22):2349-61. doi: 10.1001/jama.2009.813. PMID 19509382
- [Result] Dong H, Chen L. B7-H1 pathway and its role in the evasion of tumor immunity. J Mol Med (Berl). 2003 May;81(5):281-7. doi: 10.1007/s00109-003-0430-2. Epub 2003 Apr 30. PMID 12721664
- [Result] Chen X, Liu S, Wang L, Zhang W, Ji Y, Ma X. Clinical significance of B7-H1 (PD-L1) expression in human acute leukemia. Cancer Biol Ther. 2008 May;7(5):622-7. doi: 10.4161/cbt.7.5.5689. PMID 18756622
- [Result] Ahmadzadeh M, Johnson LA, Heemskerk B, Wunderlich JR, Dudley ME, White DE, Rosenberg SA. Tumor antigen-specific CD8 T cells infiltrating the tumor express high levels of PD-1 and are functionally impaired. Blood. 2009 Aug 20;114(8):1537-44. doi: 10.1182/blood-2008-12-195792. Epub 2009 May 7. PMID 19423728
- [Result] Gao Q, Wang XY, Qiu SJ, Yamato I, Sho M, Nakajima Y, Zhou J, Li BZ, Shi YH, Xiao YS, Xu Y, Fan J. Overexpression of PD-L1 significantly associates with tumor aggressiveness and postoperative recurrence in human hepatocellular carcinoma. Clin Cancer Res. 2009 Feb 1;15(3):971-9. doi: 10.1158/1078-0432.CCR-08-1608. PMID 19188168
- [Result] Konishi J, Yamazaki K, Azuma M, Kinoshita I, Dosaka-Akita H, Nishimura M. B7-H1 expression on non-small cell lung cancer cells and its relationship with tumor-infiltrating lymphocytes and their PD-1 expression. Clin Cancer Res. 2004 Aug 1;10(15):5094-100. doi: 10.1158/1078-0432.CCR-04-0428. PMID 15297412
- [Result] Liu J, Hamrouni A, Wolowiec D, Coiteux V, Kuliczkowski K, Hetuin D, Saudemont A, Quesnel B. Plasma cells from multiple myeloma patients express B7-H1 (PD-L1) and increase expression after stimulation with IFN-gamma and TLR ligands via a MyD88-, TRAF6-, and MEK-dependent pathway. Blood. 2007 Jul 1;110(1):296-304. doi: 10.1182/blood-2006-10-051482. Epub 2007 Mar 15. PMID 17363736
- [Result] Mumprecht S, Schurch C, Schwaller J, Solenthaler M, Ochsenbein AF. Programmed death 1 signaling on chronic myeloid leukemia-specific T cells results in T-cell exhaustion and disease progression. Blood. 2009 Aug 20;114(8):1528-36. doi: 10.1182/blood-2008-09-179697. Epub 2009 May 6. PMID 19420358
- [Result] Ghebeh H, Barhoush E, Tulbah A, Elkum N, Al-Tweigeri T, Dermime S. FOXP3+ Tregs and B7-H1+/PD-1+ T lymphocytes co-infiltrate the tumor tissues of high-risk breast cancer patients: Implication for immunotherapy. BMC Cancer. 2008 Feb 23;8:57. doi: 10.1186/1471-2407-8-57. PMID 18294387
- [Result] Hamanishi J, Mandai M, Iwasaki M, Okazaki T, Tanaka Y, Yamaguchi K, Higuchi T, Yagi H, Takakura K, Minato N, Honjo T, Fujii S. Programmed cell death 1 ligand 1 and tumor-infiltrating CD8+ T lymphocytes are prognostic factors of human ovarian cancer. Proc Natl Acad Sci U S A. 2007 Feb 27;104(9):3360-5. doi: 10.1073/pnas.0611533104. Epub 2007 Feb 21. PMID 17360651
- [Result] Freeman GJ, Long AJ, Iwai Y, Bourque K, Chernova T, Nishimura H, Fitz LJ, Malenkovich N, Okazaki T, Byrne MC, Horton HF, Fouser L, Carter L, Ling V, Bowman MR, Carreno BM, Collins M, Wood CR, Honjo T. Engagement of the PD-1 immunoinhibitory receptor by a novel B7 family member leads to negative regulation of lymphocyte activation. J Exp Med. 2000 Oct 2;192(7):1027-34. doi: 10.1084/jem.192.7.1027. PMID 11015443
- [Result] Shenghui Z, Yixiang H, Jianbo W, Kang Y, Laixi B, Yan Z, Xi X. Elevated frequencies of CD4(+) CD25(+) CD127lo regulatory T cells is associated to poor prognosis in patients with acute myeloid leukemia. Int J Cancer. 2011 Sep 15;129(6):1373-81. doi: 10.1002/ijc.25791. Epub 2011 Feb 26. PMID 21105040
- [Result] Szczepanski MJ, Szajnik M, Czystowska M, Mandapathil M, Strauss L, Welsh A, Foon KA, Whiteside TL, Boyiadzis M. Increased frequency and suppression by regulatory T cells in patients with acute myelogenous leukemia. Clin Cancer Res. 2009 May 15;15(10):3325-32. doi: 10.1158/1078-0432.CCR-08-3010. Epub 2009 May 5. PMID 19417016
- [Result] Wang X, Zheng J, Liu J, Yao J, He Y, Li X, Yu J, Yang J, Liu Z, Huang S. Increased population of CD4(+)CD25(high), regulatory T cells with their higher apoptotic and proliferating status in peripheral blood of acute myeloid leukemia patients. Eur J Haematol. 2005 Dec;75(6):468-76. doi: 10.1111/j.1600-0609.2005.00537.x. PMID 16313258
- [Result] Zhou Q, Bucher C, Munger ME, Highfill SL, Tolar J, Munn DH, Levine BL, Riddle M, June CH, Vallera DA, Weigel BJ, Blazar BR. Depletion of endogenous tumor-associated regulatory T cells improves the efficacy of adoptive cytotoxic T-cell immunotherapy in murine acute myeloid leukemia. Blood. 2009 Oct 29;114(18):3793-802. doi: 10.1182/blood-2009-03-208181. Epub 2009 Sep 1. PMID 19724059
- [Result] Zhou Q, Munger ME, Highfill SL, Tolar J, Weigel BJ, Riddle M, Sharpe AH, Vallera DA, Azuma M, Levine BL, June CH, Murphy WJ, Munn DH, Blazar BR. Program death-1 signaling and regulatory T cells collaborate to resist the function of adoptively transferred cytotoxic T lymphocytes in advanced acute myeloid leukemia. Blood. 2010 Oct 7;116(14):2484-93. doi: 10.1182/blood-2010-03-275446. Epub 2010 Jun 22. PMID 20570856
- [Result] Shvets A, Chakrabarti R, Gonzalez-Quintial R, Baccala R, Theofilopoulos AN, Prud'homme GJ. Impaired negative regulation of homeostatically proliferating T cells. Blood. 2009 Jan 15;113(3):622-5. doi: 10.1182/blood-2008-03-139964. Epub 2008 Nov 20. PMID 19023118
- [Result] Bracci L, Moschella F, Sestili P, La Sorsa V, Valentini M, Canini I, Baccarini S, Maccari S, Ramoni C, Belardelli F, Proietti E. Cyclophosphamide enhances the antitumor efficacy of adoptively transferred immune cells through the induction of cytokine expression, B-cell and T-cell homeostatic proliferation, and specific tumor infiltration. Clin Cancer Res. 2007 Jan 15;13(2 Pt 1):644-53. doi: 10.1158/1078-0432.CCR-06-1209. PMID 17255288
- [Result] Wrzesinski C, Paulos CM, Gattinoni L, Palmer DC, Kaiser A, Yu Z, Rosenberg SA, Restifo NP. Hematopoietic stem cells promote the expansion and function of adoptively transferred antitumor CD8 T cells. J Clin Invest. 2007 Feb;117(2):492-501. doi: 10.1172/JCI30414. PMID 17273561
- [Result] Wrzesinski C, Paulos CM, Kaiser A, Muranski P, Palmer DC, Gattinoni L, Yu Z, Rosenberg SA, Restifo NP. Increased intensity lymphodepletion enhances tumor treatment efficacy of adoptively transferred tumor-specific T cells. J Immunother. 2010 Jan;33(1):1-7. doi: 10.1097/CJI.0b013e3181b88ffc. PMID 19952961
- [Result] Dudley ME, Wunderlich JR, Robbins PF, Yang JC, Hwu P, Schwartzentruber DJ, Topalian SL, Sherry R, Restifo NP, Hubicki AM, Robinson MR, Raffeld M, Duray P, Seipp CA, Rogers-Freezer L, Morton KE, Mavroukakis SA, White DE, Rosenberg SA. Cancer regression and autoimmunity in patients after clonal repopulation with antitumor lymphocytes. Science. 2002 Oct 25;298(5594):850-4. doi: 10.1126/science.1076514. Epub 2002 Sep 19. PMID 12242449
- [Result] Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, Royal RE, Kammula U, White DE, Mavroukakis SA, Rogers LJ, Gracia GJ, Jones SA, Mangiameli DP, Pelletier MM, Gea-Banacloche J, Robinson MR, Berman DM, Filie AC, Abati A, Rosenberg SA. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol. 2005 Apr 1;23(10):2346-57. doi: 10.1200/JCO.2005.00.240. PMID 15800326
- [Derived] Solomon SR, Solh M, Morris LE, Holland HK, Bachier-Rodriguez L, Zhang X, Guzowski C, Jackson KC, Brown S, Bashey A. Phase 2 study of PD-1 blockade following autologous transplantation for patients with AML ineligible for allogeneic transplant. Blood Adv. 2023 Sep 26;7(18):5215-5224. doi: 10.1182/bloodadvances.2023010477. PMID 37379271

RESULTS

PARTICIPANT FLOW:
Groups:
- Lymphodepletion Plus Pembrolizumab: Fludarabine & Melphalan followed by autologous stem cell transplantation. Pembrolizumab will begin on Day +1.
  Fludarabine
  Melphalan
  Pembrolizumab
Period: Overall Study
Arm/Group | Lymphodepletion Plus Pembrolizumab
Started | 20
Completed | 15
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Lymphodepletion Plus Pembrolizumab
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 64 [26 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With 2-year Relapse Risk
Description: Hypothesis is that following lymphodepleting chemotherapy and pembrolizumab, the 2-year relapse risk will decrease to ≤35%
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lymphodepletion Plus Pembrolizumab
Number analyzed (Participants) | 20
Participants | 10

2. Secondary Outcome: Assess Safety of Pembrolizumab by Recording the Number of Participants With Treatment-related Adverse Events
Description: Assess safety of pembrolizumab in patients with AML following lymphodepleting chemotherapy
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lymphodepletion Plus Pembrolizumab
Number analyzed (Participants) | 20
Participants | 9

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Lymphodepletion Plus Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lymphodepletion Plus Pembrolizumab (N=20)
Neutropenic fever (Infections and infestations) | 7
Diarrhea (Gastrointestinal disorders) | 4
Weakness (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Failure to thrive (Musculoskeletal and connective tissue disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Mucositis (Gastrointestinal disorders) | 1
Right flank pain (Musculoskeletal and connective tissue disorders) | 1
Decreased appetite (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Non-neutropenic fever (Infections and infestations) | 5
Hypotension (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
General infection (Infections and infestations) | 2
Cytopenia (Blood and lymphatic system disorders) | 2
Radial fracture (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lymphodepletion Plus Pembrolizumab (N=20)
Cytopenias (Blood and lymphatic system disorders) | 20
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 5
Colitis (Gastrointestinal disorders) | 2
Mucositis (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Hypertension (Cardiac disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT02771197/Prot_SAP_000.pdf